CLINICAL TRIAL: NCT03935256
Title: Phase II Study of Concurrent and Sequential Carboplatin and Paclitaxel With Adjuvant Radiotherapy for High Risk Endometrial Cancer
Brief Title: Adjuvant Sequential & Concurrent CarboTaxol + Radiotherapy for High Risk Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Matthew Harkenrider, Associate Professor and Medical Director Radiation Oncology, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211704
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Endometrial Cancer
Keywords: Cancer; High Risk Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Full Dose Chemo, Reduced Dose Chemo + RT, Full Dose Chemo (Experimental): Week 1 : Cycle 1: Full Dose Carboplatin and Paclitaxel Week 4: Pelvic Radiotherapy Begins Cycle 2: Dose reduced Carboplatin and Paclitaxel Week 7 : Cycle 3: Dose reduced Carboplatin and Paclitaxel Weeks 10,13,16: Cycle 4-6: Full Dose Carboplatin and Paclitaxel
  Interventions: Drug: Carboplatin and Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin and Paclitaxel — Regimen I: Carboplatin AUC 6 & Paclitaxel 175mg/m2 given intravenously for 4 cycles during weeks 1, 10, 13, 16 Regimen II: Carboplatin AUC 2 & Paclitaxel 45mg/m2 given intravenously for 2 cycles during weeks 4 & 7 concurrent with radiotherapy
  Other Names: Paraplatin; Taxol
Radiation: Radiation Therapy — An external beam radiation dose of 45 Gy in 25 fractions is routinely prescribed to the Planning Target Volume (PTV) for postoperative radiotherapy.
  The Vaginal Brachytherapy (VBT) Boost will be delivered after the external beam radiation. Doses of 12-18 Gy in 2-3 fractions are often prescribed to the surface of the vagina to a treatment length of 3-5 cm. There is no standard dose or fractionation schedule, so this dose, fractionation, location of dose specification , and length of vagina treated will be individualized for the patient and will be at the discretion of the treating radiation oncologist.

SUMMARY:
The purpose of this trial is to evaluate the safety of sequential and concurrent carboplatin and paclitaxel with adjuvant external beam radiotherapy for locally advanced endometrial cancer. The primary objective is to assess the acute toxicities namely grade 3-4 non hematologic and grade 4 hematologic toxicities associated with the above regimen. The null hypothesis is that the unacceptable toxic response rate is ≥40%. This will be tested against a one-sided alternative that the toxicity rate is 20% or less. Simon's two-stage design was used to power this aim. In the first stage, 11 patients will be accrued. If there are 5 or more toxic responses in these 11 patients, the study will be stopped for safety reasons. Otherwise, 13 additional patients will be accrued for a total of 24 patients. Under these conditions, the probability of stopping early is 47% if the toxic response rate is truly higher than 20.0%. If this regimen is safe then its efficacy can be studied in a Phase III study.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic malignancy in the United States. Risk factors for development of endometrial cancer include increasing age, early menarche, late menopause, nulliparity, obesity, use of unopposed estrogen, and Lynch syndrome. The most common histology is endometrioid type adenocarcinoma, but less common, high-risk histologies include serous carcinoma, clear cell carcinoma, and carcinosarcoma. High risk stage I-II disease includes those with high risk histologies or any histology with multiple high risk features including deep myometrial invasion, high grade, and presence of extensive lymphovascular invasion. Locally advanced risk disease is routinely classified as Stage III-IVA. Despite treatment with adjuvant radiotherapy, chemotherapy, or combination radiotherapy and chemotherapy, relapse-free survival rates are 58-75% in modern series of GOG 258 and PORTEC-3. Therefore, there is significant need for improved therapies and optimization of combination therapy to improve these outcomes.

Standard initial management of endometrial cancer is total hysterectomy, bilateral salpingo-oophorectomy, and peritoneal washings with or without pelvic and paraaortic lymph node dissection. Endometrial cancer is surgically staged according the International Federation of Gynecologic Oncology (FIGO). Endometrioid type carcinomas most commonly present in an early stage, and several studies have established risk factors for recurrence including increasing depth of myometrial invasion, high grade, lymphovascular space invasion (LVSI), older age, greater tumor size, and increasing stage.

Historically, the rationale behind including adjuvant chemotherapy, either simultaneously with radiation therapy or sequentially, was the high rate of distant metastases despite lower pelvic failure rates with adjuvant radiation. The combination of chemotherapy and radiation therapy has additionally been shown to have greater survival compared either modality as monotherapy.

This study is designed to test the safety of adjuvant chemotherapy and radiotherapy with a novel regimen that addresses several of the hypotheses regarding the differing rate of distant metastases in GOG 258 while still using radiotherapy due to the locoregional control benefit from PORTEC-3.

To the knowledge of the investigators, no prospective study has reported on sequential and concurrent carboplatin and paclitaxel with EBRT for surgically managed endometrial cancer patients. With expeditious initiation of high dose systemic therapy and use of platinum/taxane combination chemotherapy concurrent with radiotherapy, we can address several potential hypotheses regarding the role that chemotherapy has to decrease the risk of distant metastases. Our primary objective is to assess the acute toxicities associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. If this regimen is safe, then its efficacy can be studied in a Phase III study.

This study will include high risk early stage and locally advanced endometrial cancer patients who are surgically managed with total or radical hysterectomy. Patients will be included if combination radiation therapy and chemotherapy is recommended. The most common patients to be enrolled Endometrioid type FIGO Stage I-II with high risk features, IIIC1 & IVA OR Serous Carcinoma, Clear Cell Carcinoma, Carcinosarcoma Stage I-IIIC1 & IVA

ELIGIBILITY:
Inclusion Criteria:

* Surgically managed endometrial cancer with total or radical hysterectomy with pathology of endometrioid, serous, clear cell or carcinosarcoma histologies

  * Any patient for whom combination of adjuvant radiotherapy and chemotherapy is recommended following pathology review

    * Endometrioid type FIGO Stage I-II with high risk features AND IIIC1, IVA
    * Serous Carcinoma, Clear Cell Carcinoma, Carcinosarcoma Stage I-IIIC1, IVA
* ECOG Performance Status 0-2
* No prior history of pelvic radiotherapy
* No clinical or radiographic evidence of nodal disease or distant metastases
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Patients undergoing irradiation of the para-aortic node chain
* Prior history of endometrial cancer
* Prior local radiotherapy for a pelvic malignancy
* Prior platinum or taxane based chemotherapy for any malignancy
* Patients receiving any other investigational agents
* Patients with a known malignancy with a disease free interval < 6 months prior to enrollment
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, severely symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that could limit compliance with study requirements
* Patients enrolled on a competing investigational study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicities (CTCAE v5.0) | 24 weeks
  The primary outcome will be the number of Grade 3-4 acute non-hematologic and grade 4 hematologic toxicities associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients as described in CTCAE version 5.0. These toxicities will be assess during the on treatment visits by the radiation and medical oncologist. If there are 5 or more toxic responses in the first 11 patients the study will be stopped for safety reasons.

SECONDARY OUTCOMES:
Treatment Delays | 24 weeks
  To assess the number treatment delays in scheduled therapy > 3 weeks associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients.
Chronic Toxicities (CTCAE v5.0) | 52 weeks
  To assess chronic toxicities associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients.
local control | 52 weeks
  To evaluate the disease specific outcome of local control associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.
pelvic failure-free survival | 52 weeks
  To evaluate the disease specific outcome of pelvic failure-free survival associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.
distant metastasis-free survival | 52 weeks
  To evaluate the disease specific outcome of distant metastasis-free survival associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.
disease-free survival | 52 weeks
  To evaluate the disease specific outcome of disease-free survival associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.
cause-specific survival | 52 weeks
  To evaluate the disease specific outcome of cause-specific survival associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.
overall survival | 52 weeks
  To evaluate the outcome of overall survival associated with sequential and concurrent carboplatin and paclitaxel with EBRT in the adjuvant management of endometrial cancer patients. These endpoints will be assessed clinically and radiographically.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harkenrider, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Marywood, Illinois, United States

REFERENCES:
- [Background] Bachaud JM, Fu RC, Delannes M, Izar F, Martel P, David JM, Shubinski RE, Daly NJ, Montana GS. Non-randomized comparative study of irradiation alone or in combination with surgery in stage Ib, IIa and "proximal" IIb carcinoma of the cervix. Radiother Oncol. 1991 Oct;22(2):104-10. doi: 10.1016/0167-8140(91)90005-2. PMID 1957000
- [Background] Conklin CM, Longacre TA. Endometrial stromal tumors: the new WHO classification. Adv Anat Pathol. 2014 Nov;21(6):383-93. doi: 10.1097/PAP.0000000000000046. PMID 25299308
- [Background] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Kitchener HC, Nijman HW, Kruitwagen RF, Nout RA, Verhoeven-Adema KW, Smit VT, Putter H, Creutzberg CL; PORTEC study group. Toxicity and quality of life after adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1114-1126. doi: 10.1016/S1470-2045(16)30120-6. Epub 2016 Jul 7. PMID 27397040
- [Background] Aalders J, Abeler V, Kolstad P, Onsrud M. Postoperative external irradiation and prognostic parameters in stage I endometrial carcinoma: clinical and histopathologic study of 540 patients. Obstet Gynecol. 1980 Oct;56(4):419-27. PMID 6999399
- [Background] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Background] Creutzberg CL, van Putten WL, Koper PC, Lybeert ML, Jobsen JJ, Warlam-Rodenhuis CC, De Winter KA, Lutgens LC, van den Bergh AC, van de Steen-Banasik E, Beerman H, van Lent M. Surgery and postoperative radiotherapy versus surgery alone for patients with stage-1 endometrial carcinoma: multicentre randomised trial. PORTEC Study Group. Post Operative Radiation Therapy in Endometrial Carcinoma. Lancet. 2000 Apr 22;355(9213):1404-11. doi: 10.1016/s0140-6736(00)02139-5. PMID 10791524
- [Background] Keys HM, Roberts JA, Brunetto VL, Zaino RJ, Spirtos NM, Bloss JD, Pearlman A, Maiman MA, Bell JG; Gynecologic Oncology Group. A phase III trial of surgery with or without adjunctive external pelvic radiation therapy in intermediate risk endometrial adenocarcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2004 Mar;92(3):744-51. doi: 10.1016/j.ygyno.2003.11.048. PMID 14984936
- [Background] Nout RA, Smit VT, Putter H, Jurgenliemk-Schulz IM, Jobsen JJ, Lutgens LC, van der Steen-Banasik EM, Mens JW, Slot A, Kroese MC, van Bunningen BN, Ansink AC, van Putten WL, Creutzberg CL; PORTEC Study Group. Vaginal brachytherapy versus pelvic external beam radiotherapy for patients with endometrial cancer of high-intermediate risk (PORTEC-2): an open-label, non-inferiority, randomised trial. Lancet. 2010 Mar 6;375(9717):816-23. doi: 10.1016/S0140-6736(09)62163-2. PMID 20206777
- [Background] Chino JP, Jones E, Berchuck A, Secord AA, Havrilesky LJ. The influence of radiation modality and lymph node dissection on survival in early-stage endometrial cancer. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1872-9. doi: 10.1016/j.ijrobp.2011.03.054. Epub 2011 Jun 2. PMID 21640502
- [Background] ASTEC/EN.5 Study Group; Blake P, Swart AM, Orton J, Kitchener H, Whelan T, Lukka H, Eisenhauer E, Bacon M, Tu D, Parmar MK, Amos C, Murray C, Qian W. Adjuvant external beam radiotherapy in the treatment of endometrial cancer (MRC ASTEC and NCIC CTG EN.5 randomised trials): pooled trial results, systematic review, and meta-analysis. Lancet. 2009 Jan 10;373(9658):137-46. doi: 10.1016/S0140-6736(08)61767-5. Epub 2008 Dec 16. PMID 19070891
- [Background] Bosse T, Peters EE, Creutzberg CL, Jurgenliemk-Schulz IM, Jobsen JJ, Mens JW, Lutgens LC, van der Steen-Banasik EM, Smit VT, Nout RA. Substantial lymph-vascular space invasion (LVSI) is a significant risk factor for recurrence in endometrial cancer--A pooled analysis of PORTEC 1 and 2 trials. Eur J Cancer. 2015 Sep;51(13):1742-50. doi: 10.1016/j.ejca.2015.05.015. Epub 2015 Jun 3. PMID 26049688
- [Background] Canlorbe G, Bendifallah S, Laas E, Raimond E, Graesslin O, Hudry D, Coutant C, Touboul C, Bleu G, Collinet P, Cortez A, Darai E, Ballester M. Tumor Size, an Additional Prognostic Factor to Include in Low-Risk Endometrial Cancer: Results of a French Multicenter Study. Ann Surg Oncol. 2016 Jan;23(1):171-7. doi: 10.1245/s10434-015-4583-3. Epub 2015 May 8. PMID 25952272
- [Background] Doll KM, Tseng J, Denslow SA, Fader AN, Gehrig PA. High-grade endometrial cancer: revisiting the impact of tumor size and location on outcomes. Gynecol Oncol. 2014 Jan;132(1):44-9. doi: 10.1016/j.ygyno.2013.10.023. Epub 2013 Oct 29. PMID 24183734
- [Background] Creutzberg CL, van Putten WL, Warlam-Rodenhuis CC, van den Bergh AC, de Winter KA, Koper PC, Lybeert ML, Slot A, Lutgens LC, Stenfert Kroese MC, Beerman H, van Lent M; postoperative Radiation Therapy in Endometrial Carcinoma Trial. Outcome of high-risk stage IC, grade 3, compared with stage I endometrial carcinoma patients: the Postoperative Radiation Therapy in Endometrial Carcinoma Trial. J Clin Oncol. 2004 Apr 1;22(7):1234-41. doi: 10.1200/JCO.2004.08.159. PMID 15051771
- [Background] Greven K, Winter K, Underhill K, Fontenesci J, Cooper J, Burke T. Final analysis of RTOG 9708: adjuvant postoperative irradiation combined with cisplatin/paclitaxel chemotherapy following surgery for patients with high-risk endometrial cancer. Gynecol Oncol. 2006 Oct;103(1):155-9. doi: 10.1016/j.ygyno.2006.02.007. Epub 2006 Mar 20. PMID 16545437
- [Background] Viswanathan AN, Moughan J, Miller BE, Xiao Y, Jhingran A, Portelance L, Bosch WR, Matulonis UA, Horowitz NS, Mannel RS, Souhami L, Erickson BA, Winter KA, Small W Jr, Gaffney DK. NRG Oncology/RTOG 0921: A phase 2 study of postoperative intensity-modulated radiotherapy with concurrent cisplatin and bevacizumab followed by carboplatin and paclitaxel for patients with endometrial cancer. Cancer. 2015 Jul 1;121(13):2156-63. doi: 10.1002/cncr.29337. Epub 2015 Apr 6. PMID 25847373
- [Background] Morrow CP, Bundy BN, Homesley HD, Creasman WT, Hornback NB, Kurman R, Thigpen JT. Doxorubicin as an adjuvant following surgery and radiation therapy in patients with high-risk endometrial carcinoma, stage I and occult stage II: a Gynecologic Oncology Group Study. Gynecol Oncol. 1990 Feb;36(2):166-71. doi: 10.1016/0090-8258(90)90166-i. PMID 2298404
- [Background] Fields AL, Einstein MH, Novetsky AP, Gebb J, Goldberg GL. Pilot phase II trial of radiation "sandwiched" between combination paclitaxel/platinum chemotherapy in patients with uterine papillary serous carcinoma (UPSC). Gynecol Oncol. 2008 Jan;108(1):201-6. doi: 10.1016/j.ygyno.2007.09.025. Epub 2007 Nov 8. PMID 17997145
- [Background] Hogberg T, Signorelli M, de Oliveira CF, Fossati R, Lissoni AA, Sorbe B, Andersson H, Grenman S, Lundgren C, Rosenberg P, Boman K, Tholander B, Scambia G, Reed N, Cormio G, Tognon G, Clarke J, Sawicki T, Zola P, Kristensen G. Sequential adjuvant chemotherapy and radiotherapy in endometrial cancer--results from two randomised studies. Eur J Cancer. 2010 Sep;46(13):2422-31. doi: 10.1016/j.ejca.2010.06.002. Epub 2010 Jul 7. PMID 20619634
- [Background] Small W Jr, Strauss JB, Hwang CS, Cohen L, Lurain J. Should uterine tandem applicators ever be placed without ultrasound guidance? No: a brief report and review of the literature. Int J Gynecol Cancer. 2011 Jul;21(5):941-4. doi: 10.1097/IGC.0b013e31821bca53. PMID 21697682
- [Background] Milgrom SA, Kollmeier MA, Abu-Rustum NR, Tew WP, Sonoda Y, Barakat RR, Alektiar KM. Postoperative external beam radiation therapy and concurrent cisplatin followed by carboplatin/paclitaxel for stage III (FIGO 2009) endometrial cancer. Gynecol Oncol. 2013 Sep;130(3):436-40. doi: 10.1016/j.ygyno.2013.06.024. Epub 2013 Jun 22. PMID 23800696
- [Background] Albuquerque K, Folkert M, Mayadev J, Christie A, Liotta MR, Nagel C, Sevak P, Harkenrider MM, Lea JS, Hanna RK, Small WC Jr, Miller DS, Xie XJ, Potkul RK, Elshaikh MA. Adjuvant External Radiation Impacts Outcome of Pelvis-limited Stage III Endometrial Carcinoma: A Multi-institutional Study. Am J Clin Oncol. 2018 Aug;41(8):792-796. doi: 10.1097/COC.0000000000000371. PMID 28225446
- [Background] Greven K, Winter K, Underhill K, Fontenesci J, Cooper J, Burke T; Radiation Therapy Oncology Group. Preliminary analysis of RTOG 9708: Adjuvant postoperative radiotherapy combined with cisplatin/paclitaxel chemotherapy after surgery for patients with high-risk endometrial cancer. Int J Radiat Oncol Biol Phys. 2004 May 1;59(1):168-73. doi: 10.1016/j.ijrobp.2003.10.019. PMID 15093913
- [Background] Klopp AH, Yeung AR, Deshmukh S, Gil KM, Wenzel L, Westin SN, Gifford K, Gaffney DK, Small W Jr, Thompson S, Doncals DE, Cantuaria GHC, Yaremko BP, Chang A, Kundapur V, Mohan DS, Haas ML, Kim YB, Ferguson CL, Pugh SL, Kachnic LA, Bruner DW. Patient-Reported Toxicity During Pelvic Intensity-Modulated Radiation Therapy: NRG Oncology-RTOG 1203. J Clin Oncol. 2018 Aug 20;36(24):2538-2544. doi: 10.1200/JCO.2017.77.4273. Epub 2018 Jul 10. PMID 29989857
- [Background] Mell LK, Sirak I, Wei L, Tarnawski R, Mahantshetty U, Yashar CM, McHale MT, Xu R, Honerkamp-Smith G, Carmona R, Wright M, Williamson CW, Kasaova L, Li N, Kry S, Michalski J, Bosch W, Straube W, Schwarz J, Lowenstein J, Jiang SB, Saenz CC, Plaxe S, Einck J, Khorprasert C, Koonings P, Harrison T, Shi M, Mundt AJ; INTERTECC Study Group. Bone Marrow-sparing Intensity Modulated Radiation Therapy With Concurrent Cisplatin For Stage IB-IVA Cervical Cancer: An International Multicenter Phase II Clinical Trial (INTERTECC-2). Int J Radiat Oncol Biol Phys. 2017 Mar 1;97(3):536-545. doi: 10.1016/j.ijrobp.2016.11.027. Epub 2016 Nov 23. PMID 28126303
- [Background] Small W Jr, Mell LK, Anderson P, Creutzberg C, De Los Santos J, Gaffney D, Jhingran A, Portelance L, Schefter T, Iyer R, Varia M, Winter K, Mundt AJ. Consensus guidelines for delineation of clinical target volume for intensity-modulated pelvic radiotherapy in postoperative treatment of endometrial and cervical cancer. Int J Radiat Oncol Biol Phys. 2008 Jun 1;71(2):428-34. doi: 10.1016/j.ijrobp.2007.09.042. Epub 2007 Nov 26. PMID 18037584
- [Background] Murakami N, Norihisa Y, Isohashi F, Murofushi K, Ariga T, Kato T, Inaba K, Okamoto H, Ito Y, Toita T, Itami J. Proposed definition of the vaginal cuff and paracolpium clinical target volume in postoperative uterine cervical cancer. Pract Radiat Oncol. 2016 Jan-Feb;6(1):5-11. doi: 10.1016/j.prro.2015.04.008. PMID 26767622